CLINICAL TRIAL: NCT04923464
Title: A Phase 4 Decentralized Pilot Study With Wearable Technology in Cystic Fibrosis Subjects 18 Years of Age and Older Taking Commercial Elexacaftor/Tezacaftor/Ivacaftor
Brief Title: A Decentralized Study to Evaluate Physical Activity and Cough Frequency Using Wearable Technology in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX20-445-118
Record Dates: First submitted 2021-05-20; First posted 2021-06-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ELX/TEZ/IVA: CF participants who are currently on a stable regimen of commercially available ELX/TEZ/IVA will be evaluated for the performance of wearable technology devices. Wearable devices include a wrist-worn actigraphy sensor and an ambulatory cough monitoring system.

SUMMARY:
This study will evaluate the performance of wearable technology in cystic fibrosis (CF) participants taking commercial Elexacaftor (ELX)/Tezacaftor (TEZ)/Ivacaftor (IVA) utilizing a fully decentralized trial design.

ELIGIBILITY:
Key Inclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) value greater than or equal to (≥) 30 percent predicted
* Participants with an approved CF transmembrane conductance regulator gene (CFTR) genotype according to respective regional labels

Key Exclusion Criteria:

* History of solid organ or hematological transplantation
* Non-ambulatory status

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CF taking commercial ELX/TEZ/IVA will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Compliance With Actigraphy Wearable Device Measured as Percentage of Time a Participant is Wearing the Actigraphy Wearable Device | From Day 1 up to Week 12

SECONDARY OUTCOMES:
Compliance With Cough Measurement Device Measured as Percentage of Time a Participant is Wearing the Cough Measurement Device | From Day 1 up to Week 12
Number of Steps per day and Variability in Number of Steps per day Over Time | From Day 1 up to Week 12
  Number of steps will be reported as mean and variability will be reported as standard deviation (SD).
Number of Coughs per day and Variability in Number of Coughs per day Over Time | From Day 1 up to Week 12
  Number of coughs will be reported as mean and variability will be reported as SD.
Time Spent Above Sedentary Physical Activity per day and Variability in Time Spent Above Sedentary Physical Activity per day Over Time | From Day 1 up to Week 12
  Time spent above sedentary physical activity will be reported as mean and variability will be reported as SD.
Time Spent in Moderate-to-Vigorous Physical Activity per day and Variability in Time Spent in Moderate-to-Vigorous Physical Activity per day Over Time | From Day 1 up to Week 12
  Time spent in moderate-to-vigorous physical activity will be reported as mean and variability will be reported as SD.
Time Spent in Continuous Walking Bouts per day and Variability in Time Spent in Continuous Walking Bouts per day Over Time | From Day 1 up to Week 12
  Time spent in continuous walking bouts will be reported as mean and variability will be reported as SD.
Total Activity Count per day and Variability in Total Activity Count per day Over Time | From Day 1 up to Week 12
  Total activity count will be reported as mean and variability will be reported as SD.
Best 6-Minute Effort (B6ME) and Variability in B6ME Over Time | From Day 1 up to Week 12
  B6ME will be reported as mean and variability will be reported as SD.
Sleep Efficiency and Variability in Sleep Efficiency Over Time | From Day 1 up to Week 12
  Sleep efficiency measurements will be performed using wearable technology which include a wrist-worn actigraphy sensor. Sleep efficiency will be reported as mean and variability will be reported as SD.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - National Jewish Health, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Children's Hospital of Illinois at OSF Saint Francis Medical Center, Cystic Fibrosis Center, Peoria, Illinois
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Rsearch Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Mount Sinai Beth Israel, New York, New York
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UW School of Medicine & Public Health, Madison, Wisconsin
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Devon and Exeter Hospital, Exeter
  - St. James University Hospital, Leeds
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing